CLINICAL TRIAL: NCT05464836
Title: A Phase II Study to Evaluate Safety and Efficacy of CB-103 in Combination With Venetoclax in Adolescent and Young Adult Patients With Relapsed/Refractory T-cell Acute Lymphoblastic Leukemia (T-ALL)
Brief Title: Phase II Study to Evaluate Safety and Efficacy of CB-103 With Venetoclax in Adolescent and Young Adult Patients With Relapsed/Refractory T-ALL or T-LBL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor requested termination due to internal reprioritization of resources.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0547; NCI-2022-05687 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2022-07-07; First posted 2022-07-19 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Leukemia, Lymphoblastic; Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CB-103+Venetoclax (Experimental): Control T-cell acute lymphoblastic leukemia (T-ALL) or T-cell lymphoblastic leukemia (T-LBL) in adolescent and young adult patients.
  Interventions: Drug: CB-103; Drug: Venetoclax

INTERVENTIONS:
Drug: CB-103 — Given by PO
  Other Names: Cellestia
Drug: Venetoclax — Given by PO
  Other Names: ABT-199

SUMMARY:
To learn if the combination of 2 study drugs, CB-103 and venetoclax, can help to control T-cell acute lymphoblastic leukemia (T-ALL) or T-cell lymphoblastic leukemia (T-LBL) in adolescent and young adult patients

DETAILED DESCRIPTION:
Primary Objectives:

* To characterize the safety and tolerability of CB-103 in combination with Venetoclax in adolescent (12 to 18 years) and adult (19 to 60 years) patients with relapsed/refractory T-cell acute lymphoblastic leukemia (T-ALL) and T-cell lymphoblastic lymphoma (T-LBL).
* To assess the efficacy of CB-103 in combination with venetoclax by the overall response rate (ORR), defined as complete remission (CR), plus CR with incomplete blood count recovery (CRi) [1] plus partial remission (PR) [2], in adolescent, and young adult patients with relapsed/refractory T-ALL/T-LBL.

Secondary Objectives:

* To assess whether the ORR to CB-103 in combination with Venetoclax is dependent on pre-treatment expression of Notch and/or BCL2 pathway.
* To determine the preliminary assessment of CB-103 in combination with Venetoclax by other efficacy parameters such as minimal residual disease (MRD), duration of response (DoR), overall survival (OS) and event-free survival (EFS) in adolescent and young adult patients with relapsed/refractory T-ALL/T-LBL.

Exploratory Objectives:

* To explore potential correlations of ORR to treatment and additional pharmacodynamic (PD) markers, i.e., other oncogenic pathway activations that may co-occur at the start of treatment.
* To evaluate how many patients are able to transition to Hematopoietic Stem Cell

Transplant (HSCT):

* Either in the patients achieving CR after the induction and reinduction cycles;
* Or in the patients with PR or stable disease (SD) after the induction and reinduction.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent (12 to 18 years) and adult (19 to 60 years) participants who have relapsed or refractory T-cell lymphoblastic leukemia (T-ALL) or T-Cell lymphoblastic lymphoma (T-LBL) according to 2017 WHO classification [29] and NCCN v1 2021 [30]:
* Participants must have ≥ 5% blasts in the bone marrow as assessed by morphology on standard bone marrow biopsy and aspirate or less than 5% blasts in the bone marrow in presence of extramedullary relapse, excluding isolated central nervous system (CNS) relapse. However, if an adequate bone marrow sample cannot be obtained, participants may be enrolled if there is unequivocal evidence of leukemia with ≥ 5% blasts in the peripheral blood.
* Participants are eligible independently of Notch pathway activation in the leukemic blasts:

however, a fresh marrow/blood sample must be obtained before starting the study treatment to classify the participants as being either Notch positive or negative.

* Leukemic blasts must express of at least 2 of the following immune phenotyping: CD1a, CD2, CD3, CD4, CD5, CD7, CD8, CD34, TCRαβ, TCRγδ, cyCD3
* Participants have adequate performance status (ECOG ≤2) for participants ≥16 years old, Lansky score >50 for patients <16 years old.
* Participants must be 12 to 60 years of age inclusive when signing the informed consent. For participants < 18 years of age, parent or legally authorized representative (LAR) should be willing and able to give informed consent. Non-English speaking participants are eligible for whom consent process will follow institutional guidelines.
* Participants with asymptomatic CNS disease are eligible
* Participants must have adequate organ function and laboratory results (obtained within 14 days of enrollment):

  * Direct bilirubin ≤2 x upper limit of normal (ULN).
  * Serum creatinine ≤ 1.5 x ULN; or if serum creatinine > 1.5 x ULN, then serum creatinine clearance (CrCl) ≥ 50 mL/min (estimated by Cockcroft-Gault formula).
  * Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤3 x ULN; ≤5 x ULN in case of suspected leukemic liver involvement
* Females of childbearing potential must have a negative serum or urine beta-human chorionic gonadotropin (β-HCG) pregnancy test result within 14 days prior to the first dose of study drugs and must agree to use one of the following effective contraception methods during the study and for 30 days following the last dose of study drug. Effective methods of birth control include:

  * Birth control pills, skin patches, shots, subdermal implants
  * Intrauterine devices (IUDs)
  * Condom or occlusive cap (diaphragm or cervical/vault caps) used with Spermicide
  * Abstinence
* Males agree to inform study doctor right away if their partner becomes pregnant or suspects pregnancy. While in this study and for 30 days after the last treatment the participant agrees not to donate sperm for the purposes of reproduction. He agrees to use a condom while in this study and for 30 days after the last treatment.

Exclusion Criteria:

* Mixed phenotype leukemia (excluding T-ALL with myeloid antigen expression)
* History of another primary invasive malignancy that has not been definitively treated and in remission. Participants with non-melanoma skin cancers or with carcinomas in situ are eligible regardless of the time from diagnosis (including concomitant diagnoses).
* Presence of clinically significant uncontrolled CNS pathology such as epilepsy, childhood seizure, paresis, aphasia, stroke, severe brain injuries, organic brain syndrome, or psychosis.
* Participants with a cardiac ejection fraction (as measured by either MUGA or echocardiogram) < 50% or with a history of absolute decrease in LVEF of ≥ 15 absolute percentage points are excluded.
* Medical history of cardiovascular disease such as

  * Clinically significant cardiac disease including congestive heart failure (NYHA class III or IV), arrhythmia or conduction abnormality requiring medication, or cardiomyopathy
  * Clinically uncontrolled hypertension Age Blood Pressure 12 to 13 = >120/80mmHg >13 = >140/90mmHg
  * Complete left bundle branch block
  * Right bundle branch block + left anterior hemiblock
  * Congenital long QT syndrome
  * History or presence of sustained or symptomatic ventricular tachyarrhythmia, atrial fibrillation, or clinically significant resting bradycardia (< 50 bpm)
  * Corrected QT interval using Fridericia formula (QTcF) > 450 ms for males and > 470 ms for females at the screening ECG
  * QRS ≥ 110 ms
  * History of symptomatic congestive heart failure
* Participants with uncontrolled, active infections (viral, bacterial, or fungal). Infections controlled on concurrent anti-microbial agents are acceptable. Anti-microbial prophylaxis per institutional guidelines is acceptable.
* Known active hepatitis B or C infection or known seropositivity for HIV.
* Liver cirrhosis or other active severe liver disease or suspected active alcohol abuse.
* Have conditions requiring chronic systemic (not inhaled) glucocorticoid use, such as autoimmune disease or severe asthma. Low doses of corticosteroids (10 mg prednisone equivalent a day) are permitted.
* Participants with unresolved nausea, vomiting, or diarrhea of CTCAE version 5.0, grade ˃

  1 from prior therapy.
* Participants with impairment of GI function or GI disease presence that may significantly alter the absorption of CB-103 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Have current or recurrent (within 3 months) gastrointestinal disease, have conditions requiring chronic systemic glucocorticoid use, have active graft versus host disease, or have a second primary or prior malignancy that would affect the interpretation of study results. Low doses of corticosteroids (10 mg prednisone equivalent a day) are permitted.
* Prior chemotherapy/radiotherapy/investigational therapy within 2 weeks before the start of study drugs with the following exceptions: - Up to 5 days of glucocorticoids (10 mg of dexamethasone or equivalent/day) in combination with up to 3 doses of cyclophosphamide (200 mg/m2/day) are allowed as standard pre-phase treatment up to 1 day before start of study treatment.

Cytarabine up to 2gm/m2 are also allowed as standard pre-phase treatment up to 1 day before start of study treatment.

* Mercaptopurine may be dosed up to 5 days prior to first dose of CB103
* Vinca alkaloids may be dosed up to 5 days prior to first dose of CB103
* Prophylactic intrathecal (IT) chemotherapy may be dosed up to 1 day prior to first dose of CB103

  • Females who are pregnant or lactating
* Male or female participants of childbearing potential, unwilling to use an approved, effective means of contraception in accordance with institution's standards.
* Other severe, uncontrolled acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the Investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study.
* Participants who are unable or unwilling to comply with all study requirements for clinical visits, examinations, tests, and procedures.
* Participants must be excluded if they are currently enrolled in another ongoing clinical trial with anti-cancer investigational products

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Garcia, DO, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study received IRB approval June 30, 2022 and was opened to recruitment August 12, 2024. The study was terminated by the local IRB on August 12, 2024.
Groups:
- CB-103 in Combination With Venetoclax: Treatment with CB-103 + Venetoclax in Relapsed/Refractory T-ALL or T-LBL
Period: Overall Study
Arm/Group | CB-103 in Combination With Venetoclax
Started | 2
Completed | 0
Not Completed | 2
Not completed — Progression of Disease | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | CB-103 in Combination With Venetoclax
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 20.5 [20 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of CB-103 in Combination With Venetoclax
Description: Overall response rate (ORR, including CR, CRi, and PR rate) with flow cytometric assessment of minimum residual disease (MRD)
Time Frame: Average of 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | CB-103 in Combination With Venetoclax
Number analyzed (Participants) | 2
Participants
  Progressive Disease | 1
  Stable Disease | 1

ADVERSE EVENTS:
Time Frame: Average of 3 months
Description: An an adverse event or suspected adverse reaction is considered "serious" if, in the view of either the Investigator or the sponsor, it results in any of the following outcomes:
  * Death
  * A life-threatening adverse event
  * Inpatient hospitalization or prolongation of existing hospitalization
  * A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
  * A congenital anomaly/birth defect.
Arm/Group | CB-103 in Combination With Venetoclax
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CB-103 in Combination With Venetoclax (N=2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sepsis (Infections and infestations) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CB-103 in Combination With Venetoclax (N=2)
Adbominal pain (Gastrointestinal disorders) | 1 (1)
Activated partial thromboplastin time (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (7)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchpulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Cytogalovirus infection reactivation (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Eye Redness (Eye disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Hypokalemia (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
Lung infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (General disorders) | 1 (4)
Respitory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis (Blood and lymphatic system disorders) | 1 (1)
GI Hemorrhage (Gastrointestinal disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (17)
White blood cell decreased (Investigations) | 1 (9)
Toothache (Gastrointestinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Optic nerve disorder (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT05464836/Prot_SAP_000.pdf